CLINICAL TRIAL: NCT02466763
Title: Prospective Randomized Controlled Double-blinded Study Comparing Cochlear Implantation Through a Round Window Versus Cochleostomy Approach
Brief Title: Prospective Study of Round Window Versus Cochleostomy Approach to CI Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough interest in enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew L. Carlson, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-000576
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Deafness
Keywords: round window; cochlear implants; cochleostomy
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- round window (Active Comparator): Half of the participants will be randomized to the round window technique of cochlear implant device electrode insertion. Intervention for participants randomized to the round window arm include having the round window technique used for the electrode insertion during the participant's cochlear implant surgery. Participants in this arm of the study will also have a post operative CT scan at about three months after surgery.
  Interventions: Procedure: Cochlear implant surgery
- cochleostomy (Active Comparator): Half of the participants will be randomized to the cochleostomy technique of cochlear implant device electrode insertion. For the participants randomized to the cochleostomy arm, the surgeon will use a cochleostomy technique for the electrode insertion during the participant's cochlear implant surgery. Participants in this arm of the study will also have a post operative CT scan at about three months after surgery.
  Interventions: Procedure: Cochlear implant surgery

INTERVENTIONS:
Procedure: Cochlear implant surgery — Surgical placement of a cochlear implant device.

SUMMARY:
To the investigators' knowledge, no clinical study has prospectively investigated the relationship between surgical insertion technique, intracochlear electrode location, and postoperative hearing outcomes. To this end, the investigators are conducting a multicenter prospective randomized controlled double-blinded study comparing round window and cochleostomy cochlear implant electrode insertion.

DETAILED DESCRIPTION:
Cochlear implant procedure has become the standard of care for patients with severe-to-profound sensorineural hearing loss. Successful outcomes are dependent on extrinsic and intrinsic factors. Significant predictive factors for hearing outcomes in patients with CIs have been previously reported. These include, but are not limited to, duration of deafness, level of preimplant speech recognition, pre/postlingual status, and the coupling of device electrodes. Recipient age does not appear to have a significant impact on hearing outcomes in elderly candidates.

A number of recent studies have proposed that intraoperative factors may be important determinants of electrode location and possibly of audiological outcome. Preliminary reports suggest that intracochlear electrode position- specifically, placement within the ST-is associated with improved audiological outcomes. Additionally, different surgical techniques have been proposed to minimize trauma during electrode insertion and to increase the likelihood of placement within the ST - namely round window and anteroinferior cochleostomy electrode insertion.

Currently, the best surgical approach for electrode insertion is highly debated, fueled by a lack of strong evidence to support one method over another. While a number of CI centers have begun to utilize a round window approach, many large volume centers in the United States and world wide continue to routinely employ cochleostomy electrode insertions. With an increasing number of patients being implanted with greater degrees of residual hearing, such data will become critical towards reducing intracochlear injury and optimizing patient outcomes. To the investigators' knowledge, no clinical study has prospectively investigated the relationship between surgical insertion technique, intracochlear electrode location, and postoperative hearing outcomes. To this end, the investigators are initiating a multicenter prospective randomized controlled double-blinded study comparing round window and cochleostomy cochlear implant electrode insertion.

ELIGIBILITY:
Inclusion criteria are:

* 18 years of age or older,
* less than a 10-year duration of deafness in the ear to be implanted,
* primary surgery,
* normal shaped cochleae,
* no retrocochlear pathology, and
* grossly normal cognitive function.

Exclusion criteria are:

* less than 18 years of age,
* prelingual deafness, or
* greater than 10-years duration of deafness in the ear to be implanted;
* prior otologic surgery in the implanted ear (excluding tympanostomy tube placement),
* inner ear malformation present in the ear to be implanted,
* retrocochlear pathology present in the auditory system to be implanted,
* developmental delay or known cognitive impairment, or
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-05; Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Cochlear implant electrode location after surgery | about three months post op
  a standard temporal bone CT scan will be used to show the location of the electrode in the cochlea

SECONDARY OUTCOMES:
Participant levels of speech perception | Preoperatively, and at approximately 1 month, 3 months, 6 months, and 12 months postoperatively
  standard audiometry speech perception tests will be administered
Participant levels of word recognition scores | Preoperatively, and at approximately 1 month, 3 months, 6 months, and 12 months postoperatively
  standard audiometry CNC word score test will be administered
Participant levels of sentence recognition scores | Preoperatively, and at approximately 1 month, 3 months, 6 months, and 12 months postoperatively
  standard audiometry AZBio sentence score test will be administered

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Carlson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials